CLINICAL TRIAL: NCT06736171
Title: Prescription of Robotic Exoskeletons for Ambulation Recovery Post Stroke
Brief Title: Post Stroke Ambulation Recovery Using Robotic Exoskeletons
Acronym: RERC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Karen J. Nolan, PhD, Associate Director, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-1275-24
Record Dates: First submitted 2024-12-04; First posted 2024-12-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hemiparesis After Stroke
MeSH Terms: interventions — Exoskeleton Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Stroke RE (Experimental): Participants in the stroke RE group will participate 3-4 weeks, 2-3 times a week for a total of 9 robotic exoskeleton gait training sessions provided by a trained, licensed physical therapist.
  Interventions: Device: Robotic Exoskeleton
- Stroke SOC (Active Comparator): Participants in the stroke SOC group will participate 3-4 weeks, 2-3 times a week for a total of 9 standard of care gait training sessions provided by a trained, licensed physical therapist.
  Interventions: Other: SOC

INTERVENTIONS:
Device: Robotic Exoskeleton — EksoNR, Ekso Bionics, San Rafael, CA, USA Atalante X, Wandercraft, Paris, France ReStore™, Lifeward Inc, Marlborough, MA
  Arms: Stroke RE
Other: SOC — Standard of Care
  Arms: Stroke SOC

SUMMARY:
The purpose of this research study is to evaluate and compare different robotic exoskeletons (RE) and identify which is most appropriate for gait training for each patient based off their specific needs. This will help guide clinicians in prescribing the appropriate RE for rehabilitation.

DETAILED DESCRIPTION:
This study will systematically compare various commercially available REs and aid in identifying the appropriate devices for gait training prescription in individuals post-stroke based on their deficits. The objective of this study is to evaluate and compare the four groups (3 REs and standard of care treatment) using biomechanical, functional and community participation & quality of life metrics. The robotic exoskeletons being used in this study are the AtalanteX (Wandercraft), Ekso NR (Ekso Bionics), and Restore (Lifeward).

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors 3 - 8 months from a recent stroke.
* Age: 50 - 80 years
* Unilateral hemiparesis
* Medical clearance by the Medical Director
* Be able to physically fit into the exoskeleton device: Height between 60" and 76" and weight below 220 lbs
* Patient cognitive status and ability to communicate in English must be at a level consistent with that required to participate in standard motor rehabilitation (e.g. can follow directions).
* Adequate cognitive function to give informed consent, understand the training, instructions, use investigational devices and give adequate feedback.
* Have a joint range of motion within normal functional limits for ambulation.
* Have sufficient strength to use the hemiwalker, cane or walker (etc. assistive device) while wearing the RE.
* No history of injury or pathology to the unaffected limb.
* Have an appropriate walking speed as determined by the study staff.

Exclusion Criteria:

* Any medical issue that precludes full weight-bearing and ambulation (e.g. orthopedic injuries, pain, severe spasticity).
* Skin issues that would prevent wearing the device.
* Pre-existing condition that caused exercise intolerance (documented uncontrolled hypertension, coronary artery disease, cardiac arrhythmia, or congestive heart failure).
* Hospitalization for heart attack, heart surgery, or acute heart failure within 3 months of enrollment in the study.
* Uncontrolled seizure disorder, spasticity, or joint contracture that would interfere with walking.
* Neuromuscular, neurological, or orthopedic pathologies that interfere with neuromuscular function, ambulation, or limit the range of motion of the lower limbs.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
10MWT (Aim 1) | Change from Baseline 10MWT at 4 weeks
  10 meter walk test to evaluate walking speed after stroke and in response to the intervention.
6MWT (Aim 1) | Change from Baseline 6MWT at 4 weeks
  6 minute walking test to evaluate endurance after stroke and in response to the intervention
TUG (Aim 1) | Change from Baseline TUG at 4 weeks
  Timed up and go (TUG) test to measure functional balance and walking ability after stroke and in response to the intervention.
DGI (Aim 1) | Change from Baseline DGI at 4 weeks
  Dynamic Gait Index (DGI) evaluates the ability to modify balance while walking in the presence of external demands after stroke and in response to the intervention.
Berg Balance Scale (Aim 1) | Change from Baseline Berg at 4 weeks
  Measure to assess static and dynamic balance and fall risk after stroke and in response to the intervention.
Joint Range of Motion (kinematics) (Aim 2) | Change from Baseline at 4 weeks
  Kinematics gait data will be collected using a motion capture camera system to provide biomechanical outcomes.
Temporospatial Loading (Aim 2) | Change from Baseline at 4 weeks
  Step length, timing during gait cycle, limb symmetry will be collected using instrumented gait walkway and insoles.
Balance (Aim 2) | Change from Baseline at 4 weeks
  Static and dynamic balance in standing and seated positions after stroke and in response to the intervention (using Hunova (Movendo Inc, Genova, Italy) plaform).
Survey for Community Participation (Aim 3) | Change from Baseline at 4 weeks
  The Community Participation Indicators (CPI) is a self-reported 48 item objective measure survey.
Survey for Quality of Life (Aim 3) | Change from Baseline at 4 weeks
  The SS-QOL survey assesses health-related quality of life (QOL) specific to stroke survivors with 49 items across 12 domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States